CLINICAL TRIAL: NCT02509494
Title: A Staged Phase 3 Study, Including a Double-Blinded Controlled Stage to Evaluate the Safety and Immunogenicity of Ad26.ZEBOV and MVA-BN-Filo as Candidate Prophylactic Vaccines for Ebola
Brief Title: Staged Phase 3 Study to Assess the Safety and Immunogenicity of Ebola Candidate Vaccines Ad26.ZEBOV and MVA-BN-Filo
Acronym: EBOVAC-Salone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Ministry of Health and Sanitation, Sierra Leone (Other Government); University of Sierra Leone (Other); University of Oxford (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Grameen Foundation (Other); World Vision, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR107372; VAC52150EBL3001 (Other: Janssen Vaccines & Prevention B.V.); 115854 EBOVAC1 (Other Grant/Funding Number: The Trial is financed within the IMI-2 Ebola program); 2019-000691-42 (EudraCT Number)
Record Dates: First submitted 2015-06-24; First posted 2015-07-28 (Estimated); Results first posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-06

CONDITIONS: Ebola Virus Disease
Keywords: Vaccine; Ebola; Ebola virus disease; EVD; Hemorrhagic fever; Sierra Leone; Human adenovirus serotype 26 (Ad26) encoding the Ebola virus Mayinga variant glycoprotein (Ad26.ZEBOV); Safety; Immunogenicity; Modified Vaccinia Virus Ankara - Bavarian Nordic Filo-vector; (MVA-BN Filo)
MeSH Terms: conditions — Hemorrhagic Fever, Ebola; Hemorrhagic Fevers, Viral | interventions — MenACWY

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (5):
- Stage 1: Active vaccination (Experimental): Ad26.ZEBOV will be administered as a 0.5 milliliter (mL) intramuscular (IM) injection (Dose 1); MVA-BN-Filo will be administered as a 0.5 mL IM injection (Dose 2). The booster vaccination using Ad26.ZEBOV will be administered as a 0.5 mL IM injection (2 years post Dose 1).
  Interventions: Biological: Ad26.ZEBOV; Biological: MVA-BN-Filo
- Stage 2: Active vaccination (Experimental): Ad26.ZEBOV will be administered as a 0.5 mL IM injection (Dose 1); MVA-BN-Filo will be administered as a 0.5 mL IM injection (Dose 2).
  Interventions: Biological: Ad26.ZEBOV; Biological: MVA-BN-Filo
- Stage 2: Active vaccination for children (Experimental): Ad26.ZEBOV will be administered as a 0.5 mL IM injection (Dose 1); MVA-BN-Filo will be administered as a 0.5 mL IM injection (Dose 2). Children aged less than 2 years at randomization will receive a booster dose of vaccination at 3 months post Dose 2 with Placebo.
  Interventions: Biological: Ad26.ZEBOV; Biological: MVA-BN-Filo
- Stage 2: Control vaccination (Active Comparator): MenACWY will be administered as a 0.5 mL IM injection on Day 1 (Dose 1) and placebo on Day 57 (Dose 2).
  Interventions: Biological: MenACWY; Biological: Placebo
- Stage 2: Control vaccination for children (Active Comparator): MenACWY will be administered as a 0.5 mL IM injection on Day 1 (Dose 1) and placebo on Day 57 (Dose 2). Children aged less than 2 years at randomization will receive a booster dose of MenACWY vaccination at 3 months post Dose 2 with MenACWY.
  Interventions: Biological: MenACWY; Biological: Placebo

INTERVENTIONS:
Biological: Ad26.ZEBOV — Ebola Zaire vaccine, replication incompetent vaccine, sterile suspension of 0.5 milliliter (mL) intramuscular (IM) injection of 5*10^10 viral particles.
  Arms: Stage 1: Active vaccination; Stage 2: Active vaccination; Stage 2: Active vaccination for children
Biological: MVA-BN-Filo — MVA-BN-Filo- is a non-replicating vaccine, 0.5 mL IM injection of 1*10^8 Infectious Unit (Inf. U.).
  Arms: Stage 1: Active vaccination; Stage 2: Active vaccination; Stage 2: Active vaccination for children
Biological: MenACWY — MenACWY is a WHO-prequalified Meningococcal Group A, C, W135 and Y conjugate vaccine.
  Arms: Stage 2: Control vaccination; Stage 2: Control vaccination for children
Biological: Placebo — 0.9% saline for injection.
  Arms: Stage 2: Control vaccination; Stage 2: Control vaccination for children

SUMMARY:
The purpose of this study is the evaluation of the safety and immunogenicity of two candidate Ebola vaccines Ad26.ZEBOV and MVA-BN-Filo, in a 2-dose heterologous regimen.

DETAILED DESCRIPTION:
This is staged Phase 3 study to gather information on the safety and immunogenicity of a 2-dose heterologous regimen. In this regimen, Ad26.ZEBOV will be administered as a Dose 1 vaccination followed by the candidate vaccine MVA-BN-Filo (Dose 2 56 days later) and a booster dose of A26.ZEBOV will be administered 2 years post Dose 1 vaccination to participants in Stage 1 who consent to this. The study will take place in Sierra Leone and will consist of a screening phase, an active phase (vaccination) and a follow-up phase. The active phase of the study will be conducted initially in two stages. In the first stage approximately 40 adults aged 18 years or older will be vaccinated to gain information about the safety and immunogenicity of the 2-dose heterologous vaccine regimen. In stage 2 a larger group of approximately 976 individuals will be vaccinated to further evaluate the safety and immunogenicity of the 2 dose heterologous vaccine regimen across different age groups. In this stage, children aged 1 year or older, adolescents and adults will be included. Solicited local and systemic adverse events will be collected until 7 days after the Dose 1 and Dose 2 vaccination. Unsolicited adverse events will be collected from signing of the informed consent form (ICF) onwards until 56 days after the Dose 2 vaccination in Stage 1 and then again from the day of the booster vaccination until 28 days after the booster vaccination, and until 28 days after each vaccination in stage 2. Serious adverse events will be collected from signing of the ICF onwards until 12 and 36 months after the Dose 1 vaccination in Stage 2 and Stage 1, respectively. These data will be reviewed by an independent data monitoring committee (IDMC) to assess whether initiation of vaccination in the next stage or age group can be provided. Safety evaluations will include assessment of adverse events, which will be monitored throughout the study. Participants in Stage 2 will be followed up for safety and immunogenicity until 12 months (children and adolescents) or 24 months (adults) after the Dose 1 vaccination. Participants in Stage 1 will be followed up for safety and immunogenicity until 36 months after the Dose 1 vaccination or until 1 year after the booster vaccination.

ELIGIBILITY:
Inclusion Criteria Stage 1 and 2:

* Documented community engagement from community leader and a signed inform consent form (ICF) from each participant must be available
* Participant Stage 1 must be 18 years or older at screening and be resident in selected study community with no intention to move from study area within the next 5 months
* Participant must be healthy with no abnormalities in laboratory screening tests within 28 days before Dose 1 vaccination
* Female participants of childbearing potential must use adequate birth control measures and must have a negative pregnancy test at screening and immediately prior to each study vaccination
* Participant must pass the test of understanding (TOU)

Additional Inclusion criteria Stage 2:

* One year or older at screening (children of enrolled parents are eligible)
* Parent/legal guardian (for children) must pass the TOU before signing the ICF
* Subjects aged 7 years and older will be asked to give positive assent in the presence of a witness

Exclusion Criteria:

* Diagnosed with EVD or under quarantine/exposed to Ebola or body temperature equal of >= 38 degree Celsius (fever)
* Having an acute illness (mild in nature that can be treated at home) or any clinically significant acute/chronic medical condition or having a decreased number of red blood cells/hemoglobin in the blood (anemia)
* Previously participated in another Ebola interventional study or received any Ad26/MVA-based candidate vaccine
* Vaccinated with live attenuated vaccines within 30 days or with inactivated vaccines 15 days before Dose 1 vaccination
* Treated with an immunosuppressive drug at the time of screening

Additional exclusion criteria:

- Children up to 5 years of age with severe malnutrition (underweight or Z-score weight <2)

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1023 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (1):
- Freetown, Sierra Leone

REFERENCES:
- [Derived] Barry H, Lhomme E, Surenaud M, Nouctara M, Robinson C, Bockstal V, Valea I, Somda S, Tinto H, Meda N, Greenwood B, Thiebaut R, Lacabaratz C. Helminth exposure and immune response to the two-dose heterologous Ad26.ZEBOV, MVA-BN-Filo Ebola vaccine regimen. PLoS Negl Trop Dis. 2024 Apr 11;18(4):e0011500. doi: 10.1371/journal.pntd.0011500. eCollection 2024 Apr. PMID 38603720
- [Derived] Manno D, Patterson C, Drammeh A, Tetteh K, Kroma MT, Otieno GT, Lawal BJ, Soremekun S, Ayieko P, Gaddah A, Kamara AB, Baiden F, Afolabi MO, Tindanbil D, Owusu-Kyei K, Ishola D, Deen GF, Keshinro B, Njie Y, Samai M, Lowe B, Robinson C, Leigh B, Drakeley C, Greenwood B, Watson-Jones D. The Effect of Previous Exposure to Malaria Infection and Clinical Malaria Episodes on the Immune Response to the Two-Dose Ad26.ZEBOV, MVA-BN-Filo Ebola Vaccine Regimen. Vaccines (Basel). 2023 Aug 2;11(8):1317. doi: 10.3390/vaccines11081317. PMID 37631885
- [Derived] Ishola D, Manno D, Afolabi MO, Keshinro B, Bockstal V, Rogers B, Owusu-Kyei K, Serry-Bangura A, Swaray I, Lowe B, Kowuor D, Baiden F, Mooney T, Smout E, Kohn B, Otieno GT, Jusu M, Foster J, Samai M, Deen GF, Larson H, Lees S, Goldstein N, Gallagher KE, Gaddah A, Heerwegh D, Callendret B, Luhn K, Robinson C, Leyssen M, Greenwood B, Douoguih M, Leigh B, Watson-Jones D; EBL3001 study group. Safety and long-term immunogenicity of the two-dose heterologous Ad26.ZEBOV and MVA-BN-Filo Ebola vaccine regimen in adults in Sierra Leone: a combined open-label, non-randomised stage 1, and a randomised, double-blind, controlled stage 2 trial. Lancet Infect Dis. 2022 Jan;22(1):97-109. doi: 10.1016/S1473-3099(21)00125-0. Epub 2021 Sep 13. PMID 34529963
- [Derived] Afolabi MO, Ishola D, Manno D, Keshinro B, Bockstal V, Rogers B, Owusu-Kyei K, Serry-Bangura A, Swaray I, Lowe B, Kowuor D, Baiden F, Mooney T, Smout E, Kohn B, Otieno GT, Jusu M, Foster J, Samai M, Deen GF, Larson H, Lees S, Goldstein N, Gallagher KE, Gaddah A, Heerwegh D, Callendret B, Luhn K, Robinson C, Greenwood B, Leyssen M, Douoguih M, Leigh B, Watson-Jones D; EBL3001 study group. Safety and immunogenicity of the two-dose heterologous Ad26.ZEBOV and MVA-BN-Filo Ebola vaccine regimen in children in Sierra Leone: a randomised, double-blind, controlled trial. Lancet Infect Dis. 2022 Jan;22(1):110-122. doi: 10.1016/S1473-3099(21)00128-6. Epub 2021 Sep 13. PMID 34529962
- [Derived] Mooney T, Smout E, Leigh B, Greenwood B, Enria L, Ishola D, Manno D, Samai M, Douoguih M, Watson-Jones D. EBOVAC-Salone: Lessons learned from implementing an Ebola vaccine trial in an Ebola-affected country. Clin Trials. 2018 Oct;15(5):436-443. doi: 10.1177/1740774518780678. Epub 2018 Jun 12. PMID 29895178

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 1023 participants who signed informed consent form, only 1018 participants were randomized and received study treatment and were included in the analysis.
Groups:
- Stage 1 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo (Ad26.ZEBOV): Participants with >=18 years of age (adults) received Ad26.ZEBOV 5*10^10 viral particles (vp) intramuscular (IM) injection as Dose 1 on Day 1 followed by IM injection of MVA-BN-Filo 1*10^8 infectious units (Inf.U) as Dose 2 on Day 57. Participants received a third vaccination with Ad26.ZEBOV 5*10^10 vp as a booster dose 2 years post dose 1 (Day 731).
- Stage 2 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo: Participants with >=18 years of age (adults) received Ad26.ZEBOV 5*10^10 vp IM injection as Dose 1 on Day 1, followed by IM injection of MVA-BN-filo 1*10^8 Inf.U as Dose 2 on Day 57.
- Stage 2 (>=18 Years): MenACWY, Placebo: Participants with >=18 years of age (adults) received MenACWY 0.5 milliliter (mL) IM injection as Dose 1 on Day 1, followed by IM injection of placebo on Day 57.
- Stage 2 (12-17 Years): Ad26.ZEBOV, MVA-BN-Filo: Participants with 12-17 years of age received Ad26.ZEBOV 5*10^10 vp IM injection as Dose 1 on Day 1, followed by IM injection of MVA-BN-filo 1*10^8 Inf.U as dose 2 on Day 57.
- Stage 2 (12-17 Years): MenACWY, Placebo: Participants with 12-17 years of age received MenACWY 0.5 mL IM injection as Dose 1 on Day 1, followed by IM injection of placebo on Day 57.
- Stage 2 (4-11 Years): Ad26.ZEBOV, MVA-BN-Filo: Participants with 4-11 years of age received Ad26.ZEBOV 5*10^10 vp IM injection as Dose 1 on Day 1 followed by IM injection of MVA-BN-Filo 1*10^8 Inf.U as Dose 2 on Day 57.
- Stage 2 (4-11 Years): MenACWY, Placebo: Participants with 4-11 years of age received MenACWY 0.5 mL IM injection as Dose 1 on Day 1, followed by IM injection of placebo on Day 57.
- Stage 2 (1-3 Years): Ad26.ZEBOV, MVA-BN-Filo: Participants with 1-3 years of age received Ad26.ZEBOV 5*10^10 vp IM injection as Dose 1 on Day 1, followed by IM injection of MVA-BN-filo 1*10^8 inf.U as Dose 2 on Day 57, and placebo on Day 156. Third dose (placebo) is only for children less than two years old who reconsented.
- Stage 2 (1-3 Years): MenACWY, Placebo: Participants with 1-3 years of age received MenACWY 0.5 mL IM injection as Dose 1 on Day 1, followed by IM injection of placebo on Day 57 and then IM injection of MenACWY 0.5 mL on Day 156. Third dose (MenACWY) is only for children less than two years old who reconsented.
Period: Overall Study
Arm/Group | Stage 1 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo (Ad26.ZEBOV) | Stage 2 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (>=18 Years): MenACWY, Placebo | Stage 2 (12-17 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (12-17 Years): MenACWY, Placebo | Stage 2 (4-11 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (4-11 Years): MenACWY, Placebo | Stage 2 (1-3 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (1-3 Years): MenACWY, Placebo
Started | 43 | 298 | 102 | 143 | 48 | 144 | 48 | 144 | 48
Completed | 28 | 217 | 64 | 132 | 43 | 133 | 45 | 137 | 46
Not Completed | 15 | 81 | 38 | 11 | 5 | 11 | 3 | 7 | 2
Not completed — Lost to Follow-up | 8 | 47 | 19 | 6 | 3 | 3 | 1 | 3 | 1
Not completed — Physician Decision | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 17 | 7 | 5 | 0 | 6 | 1 | 2 | 1
Not completed — Death | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 4 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-Compliance With Study Drug | 1 | 11 | 7 | 0 | 1 | 2 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo (Ad26.ZEBOV) | Stage 2 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (>=18 Years): MenACWY, Placebo | Stage 2 (12-17 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (12-17 Years): MenACWY, Placebo | Stage 2 (4-11 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (4-11 Years): MenACWY, Placebo | Stage 2 (1-3 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (1-3 Years): MenACWY, Placebo | Total
Number analyzed (Participants) | 43 | 298 | 102 | 143 | 48 | 144 | 48 | 144 | 48 | 1018
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (9.87) | 27.5 (10.46) | 29.6 (11.6) | 14.2 (1.58) | 14 (1.58) | 7.7 (1.88) | 7.9 (1.96) | 1.9 (0.79) | 1.9 (0.76) | 16.6 (12.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 50 | 22 | 69 | 21 | 73 | 26 | 67 | 21 | 350
  Male | 42 | 248 | 80 | 74 | 27 | 71 | 22 | 77 | 27 | 668
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 43 | 298 | 102 | 143 | 47 | 144 | 48 | 144 | 48 | 1017
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 43 | 297 | 102 | 142 | 47 | 144 | 47 | 144 | 48 | 1014
  White | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 4
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  SIERRA LEONE | 43 | 298 | 102 | 143 | 48 | 144 | 48 | 144 | 48 | 1018

OUTCOME MEASURES:

1. Primary Outcome: Stages 1 and 2: Number of Participants With Solicited Local Adverse Events (AEs) (Day 8)
Description: Number of participants with solicited local AEs were reported. Solicited local AEs were pre-defined local (at the injection site) AEs for which participants were specifically questioned and which were noted by participants in their diary for 7 days post vaccination. Solicited local AEs were: injection site pain/tenderness, erythema, induration/swelling, itching at the vaccination site.
Time Frame: 7 days post dose 1 (Day 8)
Population: The Full Analysis Set (FAS) included all participants who received at least one dose of study vaccine (Ad26.ZEBOV, MVA-BN-Filo or control), regardless of the occurrence of protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo (Ad26.ZEBOV) | Stage 2 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (>=18 Years): MenACWY, Placebo | Stage 2 (12-17 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (12-17 Years): MenACWY, Placebo | Stage 2 (4-11 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (4-11 Years): MenACWY, Placebo | Stage 2 (1-3 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (1-3 Years): MenACWY, Placebo
Number analyzed (Participants) | 43 | 298 | 102 | 143 | 48 | 144 | 48 | 144 | 48
Participants | 12 | 51 | 17 | 14 | 3 | 30 | 2 | 21 | 5

2. Primary Outcome: Stages 1 and 2: Number of Participants With Solicited Local AEs (Day 64)
Description: as for outcome 1
Time Frame: 7 days post dose 2 (Day 64)
Population: The FAS included all participants who received at least one dose of study vaccine (Ad26.ZEBOV, MVA-BN-Filo or control), regardless of the occurrence of protocol deviations. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo (Ad26.ZEBOV) | Stage 2 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (>=18 Years): MenACWY, Placebo | Stage 2 (12-17 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (12-17 Years): MenACWY, Placebo | Stage 2 (4-11 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (4-11 Years): MenACWY, Placebo | Stage 2 (1-3 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (1-3 Years): MenACWY, Placebo
Number analyzed (Participants) | 43 | 246 | 86 | 142 | 46 | 143 | 48 | 143 | 48
Participants | 6 | 58 | 8 | 21 | 1 | 22 | 5 | 7 | 0

3. Primary Outcome: Stage 1: Number of Participants With Solicited Local AEs (Day 738)
Description: as for outcome 1
Time Frame: 7 days post dose 3 (Day 738)
Population: The FAS included all participants who received booster dose with Ad26.ZEBOV, regardless of the occurrence of protocol deviations. This outcome measure was only planned for participants who received booster vaccination with Ad26.ZEBOV hence other arms are not reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo (Ad26.ZEBOV)
Number analyzed (Participants) | 29
Participants | 5

4. Primary Outcome: Stages 1 and 2: Number of Participants With Solicited Systemic AEs (Day 8)
Description: Number of participants with solicited systemic AEs were reported. Solicited systemic AEs included body temperature, vomiting, reduced activity, somnolence, fatigue, irritability/fussiness/crying/screaming, and loss of appetite (for preverbal children/infants) and body temperature, nausea/vomiting, fatigue/malaise, muscle pain, chills, joint pain and headache (for young children, adolescents, and adults).
Time Frame: 7 days post dose 1 (Day 8)
Population: The FAS included all participants who received at least one dose of study vaccine (Ad26.ZEBOV, MVA-BN-Filo or control), regardless of the occurrence of protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo (Ad26.ZEBOV) | Stage 2 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (>=18 Years): MenACWY, Placebo | Stage 2 (12-17 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (12-17 Years): MenACWY, Placebo | Stage 2 (4-11 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (4-11 Years): MenACWY, Placebo | Stage 2 (1-3 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (1-3 Years): MenACWY, Placebo
Number analyzed (Participants) | 43 | 298 | 102 | 143 | 48 | 144 | 48 | 144 | 48
Participants | 18 | 161 | 51 | 52 | 14 | 45 | 15 | 36 | 12

5. Primary Outcome: Stages 1 and 2: Number of Participants With Solicited Systemic AEs (Day 64)
Description: as for outcome 4
Time Frame: 7 days post dose 2 (Day 64)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo (Ad26.ZEBOV) | Stage 2 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (>=18 Years): MenACWY, Placebo | Stage 2 (12-17 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (12-17 Years): MenACWY, Placebo | Stage 2 (4-11 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (4-11 Years): MenACWY, Placebo | Stage 2 (1-3 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (1-3 Years): MenACWY, Placebo
Number analyzed (Participants) | 43 | 246 | 86 | 142 | 46 | 143 | 48 | 143 | 48
Participants | 17 | 107 | 39 | 26 | 6 | 27 | 8 | 23 | 14

6. Primary Outcome: Stage 1: Number of Participants With Solicited Systemic AEs (Day 738)
Description: as for outcome 4
Time Frame: 7 days post dose 3 (Up to Day 738)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo (Ad26.ZEBOV)
Number analyzed (Participants) | 29
Participants | 9

7. Primary Outcome: Stages 1: Number of Participants With Serious Adverse Events (SAEs)
Description: Number of Participants with SAEs were reported. SAE is any untoward medical occurrence that at any dose may result in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product.
Time Frame: Up to 36 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo (Ad26.ZEBOV)
Number analyzed (Participants) | 43
Participants | 3

8. Primary Outcome: Stages 2: Number of Participants With SAEs
Description: as for outcome 7
Time Frame: Up to 24 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (>=18 Years): MenACWY, Placebo | Stage 2 (12-17 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (12-17 Years): MenACWY, Placebo | Stage 2 (4-11 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (4-11 Years): MenACWY, Placebo | Stage 2 (1-3 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (1-3 Years): MenACWY, Placebo
Number analyzed (Participants) | 298 | 102 | 143 | 48 | 144 | 48 | 144 | 48
Participants | 16 | 4 | 0 | 1 | 5 | 0 | 15 | 3

9. Primary Outcome: Stage 1: Number of Participants With Unsolicited AEs (Day 759)
Description: Number of participants with unsolicited AEs were reported. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days post booster dose (Day 759)
Population: The FAS included all participants who received booster dose with Ad26.ZEBOV, regardless of the occurrence of protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo (Ad26.ZEBOV)
Number analyzed (Participants) | 29
Participants | 5

10. Primary Outcome: Stage 1: Number of Participants With Unsolicited AEs (Day 29)
Description: as for outcome 9
Time Frame: 28 days post dose 1 (Day 29)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo (Ad26.ZEBOV)
Number analyzed (Participants) | 43
Participants | 17

11. Primary Outcome: Stage 2: Number of Participants With Unsolicited AEs (Day 29)
Description: as for outcome 9
Time Frame: 28 days post dose 1 (Day 29)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (>=18 Years): MenACWY, Placebo | Stage 2 (12-17 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (12-17 Years): MenACWY, Placebo | Stage 2 (4-11 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (4-11 Years): MenACWY, Placebo | Stage 2 (1-3 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (1-3 Years): MenACWY, Placebo
Number analyzed (Participants) | 298 | 102 | 143 | 48 | 144 | 48 | 144 | 48
Participants | 198 | 65 | 54 | 20 | 60 | 18 | 88 | 28

12. Primary Outcome: Stage 1: Number of Participants With Unsolicited AEs (Day 85)
Description: as for outcome 9
Time Frame: 28 days post dose 2 (Day 85)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo (Ad26.ZEBOV)
Number analyzed (Participants) | 43
Participants | 17

13. Primary Outcome: Stage 2: Number of Participants With Unsolicited AEs (Day 85)
Description: as for outcome 9
Time Frame: 28 days post dose 2 (Day 85)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (>=18 Years): MenACWY, Placebo | Stage 2 (12-17 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (12-17 Years): MenACWY, Placebo | Stage 2 (4-11 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (4-11 Years): MenACWY, Placebo | Stage 2 (1-3 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (1-3 Years): MenACWY, Placebo
Number analyzed (Participants) | 246 | 86 | 142 | 46 | 143 | 48 | 143 | 48
Participants | 145 | 48 | 49 | 13 | 46 | 13 | 92 | 31

14. Primary Outcome: Stage 1: Number of Participants With Deaths
Description: Number of participants with deaths were reported.
Time Frame: Up to 36 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo (Ad26.ZEBOV)
Number analyzed (Participants) | 43
Participants | 0

15. Primary Outcome: Stage 2: Number of Participants With Deaths (Children and Adolescents)
Description: Number of participants (children and adolescents) with deaths were reported.
Time Frame: Up to 12 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2 (12-17 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (12-17 Years): MenACWY, Placebo | Stage 2 (4-11 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (4-11 Years): MenACWY, Placebo | Stage 2 (1-3 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (1-3 Years): MenACWY, Placebo
Number analyzed (Participants) | 143 | 48 | 144 | 48 | 144 | 44
Participants | 0 | 1 | 0 | 0 | 1 | 0

16. Primary Outcome: Stage 2: Number of Participants With Deaths (Adults)
Description: Number of participants (adults) with deaths were reported.
Time Frame: Up to 24 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (>=18 Years): MenACWY, Placebo
Number analyzed (Participants) | 298 | 102
Participants | 1 | 0

17. Primary Outcome: Stage 1: Number of Participants With Immediate Reportable Event (IREs)
Description: Number of participants with IREs were reported. The following list of neuroinflammatory disorders are categorized as IREs: Cranial nerve disorders, including paralyses/paresis, optic neuritis, multiple sclerosis, transverse myelitis, guillain-Barré syndrome, acute disseminated encephalomyelitis, including site specific variants, myasthenia gravis and Lambert-Eaton myasthenic syndrome, immune-mediated peripheral neuropathies and plexopathies, narcolepsy, isolated paresthesia of greater than (>) 7 days duration.
Time Frame: Up to 36 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo (Ad26.ZEBOV)
Number analyzed (Participants) | 43
Participants | 0

18. Primary Outcome: Stage 2: Number of Participants With IREs (Children and Adolescents)
Description: Number of participants (children and adolescents) with IREs were reported. The following list of neuroinflammatory disorders are categorized as IREs: Cranial nerve disorders, including paralyses/paresis, optic neuritis, multiple sclerosis, transverse myelitis, guillain-Barré syndrome, acute disseminated encephalomyelitis, including site specific variants, myasthenia gravis and Lambert-Eaton myasthenic syndrome, immune-mediated peripheral neuropathies and plexopathies, narcolepsy, isolated paresthesia of greater than (>) 7 days duration.
Time Frame: Up to 12 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2 (12-17 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (12-17 Years): MenACWY, Placebo | Stage 2 (4-11 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (4-11 Years): MenACWY, Placebo | Stage 2 (1-3 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (1-3 Years): MenACWY, Placebo
Number analyzed (Participants) | 143 | 48 | 144 | 48 | 144 | 48
Participants | 0 | 0 | 0 | 0 | 0 | 0

19. Primary Outcome: Stage 2: Number of Participants With IREs (Adults)
Description: Number of participants (adults) with IREs were reported. The following list of neuroinflammatory disorders are categorized as IREs: Cranial nerve disorders, including paralyses/paresis, optic neuritis, multiple sclerosis, transverse myelitis, guillain-Barré syndrome, acute disseminated encephalomyelitis, including site specific variants, myasthenia gravis and Lambert-Eaton myasthenic syndrome, immune-mediated peripheral neuropathies and plexopathies, narcolepsy, isolated paresthesia of greater than (>) 7 days duration.
Time Frame: Up to 24 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (>=18 Years): MenACWY, Placebo
Number analyzed (Participants) | 298 | 102
Participants | 0 | 0

20. Secondary Outcome: Stages 1 and 2: Geometric Mean Concentrations (GMCs) of Binding Antibody Levels Against Ebola Virus Glycoprotein (EBOV GP) Measured Using Enzyme-linked Immunosorbent Assay (ELISA)
Description: GMCs of antibodies binding to EBOV GP using ELISA were reported and were measured in ELISA units per milliliter (EU/mL). Serum samples were collected for analysis of binding antibodies against EBOV GP using ELISA to determine humoral responses following vaccination. For ELISA binding antibody responses, values below the lower limit of quantification (LLOQ) (36.11 ELISA units/mL).
Time Frame: 21 days post-dose 2 (Day 78)
Population: The per protocol analysis set included all randomized and vaccinated participants, who received both the prime and boost vaccinations had at least 1 post-vaccination evaluable immunogenicity sample, and had no major protocol violations influencing the immune response. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units/mL
Arm/Group | Stage 1 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo (Ad26.ZEBOV) | Stage 2 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (>=18 Years): MenACWY, Placebo | Stage 2 (12-17 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (12-17 Years): MenACWY, Placebo | Stage 2 (4-11 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (4-11 Years): MenACWY, Placebo | Stage 2 (1-3 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (1-3 Years): MenACWY, Placebo
Number analyzed (Participants) | 42 | 182 | 62 | 134 | 46 | 124 | 43 | 124 | 38
ELISA units/mL | 4784 [3736 to 6125] | 3810 [3312 to 4383] | 50 [NA to 70] — Here, 'NA' signifies that lower limit of calculated 95% CI was less than LLOQ. | 9929 [8172 to 12064] | 74 [48 to 114] | 10212 [8419 to 12388] | 42 [NA to 60] — Here, 'NA' signifies that lower limit of calculated 95% CI was less than LLOQ. | 22568 [18426 to 27642] | NA [NA to 38] — Here, 'NA' signifies that geometric mean and lower limit of calculated 95% CI was less than LLOQ.

ADVERSE EVENTS:
Time Frame: Stage 1: Up to 36 months, Stage 2 (Children and Adolescents): Up to 12 months, Stage 2 (Adults): Up to 24 months
Description: The Full Analysis Set (FAS) included all participants who received at least one dose of study vaccine (Ad26.ZEBOV, MVA-BN-Filo or control), regardless of the occurrence of protocol deviations.
Arm/Group | Stage 1 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo (Ad26.ZEBOV) | Stage 2 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (>=18 Years): MenACWY, Placebo | Stage 2 (12-17 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (12-17 Years): MenACWY, Placebo | Stage 2 (4-11 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (4-11 Years): MenACWY, Placebo | Stage 2 (1-3 Years): Ad26.ZEBOV, MVA-BN-Filo | Stage 2 (1-3 Years): MenACWY, Placebo
All-Cause Mortality (participants affected / at risk) | 0/43 | 1/298 | 0/102 | 0/143 | 1/48 | 0/144 | 0/48 | 1/144 | 0/48
Serious Adverse Events (participants affected / at risk) | 3/43 | 16/298 | 4/102 | 0/143 | 1/48 | 5/144 | 0/48 | 15/144 | 3/48
Other Adverse Events (participants affected / at risk) | 22/43 | 194/298 | 63/102 | 56/143 | 18/48 | 69/144 | 21/48 | 108/144 | 38/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo (Ad26.ZEBOV) (N=43) | Stage 2 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo (N=298) | Stage 2 (>=18 Years): MenACWY, Placebo (N=102) | Stage 2 (12-17 Years): Ad26.ZEBOV, MVA-BN-Filo (N=143) | Stage 2 (12-17 Years): MenACWY, Placebo (N=48) | Stage 2 (4-11 Years): Ad26.ZEBOV, MVA-BN-Filo (N=144) | Stage 2 (4-11 Years): MenACWY, Placebo (N=48) | Stage 2 (1-3 Years): Ad26.ZEBOV, MVA-BN-Filo (N=144) | Stage 2 (1-3 Years): MenACWY, Placebo (N=48)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 0
Anaemia of Pregnancy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinal Detachment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peptic Ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chorioretinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Helminthic Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaria (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 14 | 2
Meningitis Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Orchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis Chronic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Postoperative Wound Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 6 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Typhoid Fever (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abortion Induced Incomplete (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multiple Injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Open Globe Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abortion Threatened (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage in Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Placenta Praevia (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Premature Labour (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal Haematoma (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypovolaemic Shock (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo (Ad26.ZEBOV) (N=43) | Stage 2 (>=18 Years): Ad26.ZEBOV, MVA-BN-Filo (N=298) | Stage 2 (>=18 Years): MenACWY, Placebo (N=102) | Stage 2 (12-17 Years): Ad26.ZEBOV, MVA-BN-Filo (N=143) | Stage 2 (12-17 Years): MenACWY, Placebo (N=48) | Stage 2 (4-11 Years): Ad26.ZEBOV, MVA-BN-Filo (N=144) | Stage 2 (4-11 Years): MenACWY, Placebo (N=48) | Stage 2 (1-3 Years): Ad26.ZEBOV, MVA-BN-Filo (N=144) | Stage 2 (1-3 Years): MenACWY, Placebo (N=48)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 1 | 3 | 6 | 4 | 13 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 8 | 3
Peptic Ulcer (Gastrointestinal disorders) | 0 | 15 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 3 | 16 | 10 | 3 | 1 | 0 | 1 | 0 | 0
Furuncle (Infections and infestations) | 6 | 11 | 3 | 2 | 1 | 1 | 2 | 6 | 3
Gastroenteritis (Infections and infestations) | 1 | 10 | 2 | 1 | 0 | 3 | 2 | 7 | 5
Malaria (Infections and infestations) | 6 | 123 | 40 | 35 | 9 | 50 | 14 | 81 | 26
Nasopharyngitis (Infections and infestations) | 0 | 21 | 5 | 1 | 0 | 5 | 0 | 6 | 5
Respiratory Tract Infection (Infections and infestations) | 2 | 15 | 4 | 6 | 2 | 4 | 4 | 17 | 5
Tinea Capitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 3
Typhoid Fever (Infections and infestations) | 1 | 14 | 9 | 0 | 0 | 1 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 16 | 8 | 3 | 1 | 9 | 4 | 26 | 9
Haemoglobin Decreased (Investigations) | 0 | 7 | 2 | 8 | 5 | 3 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 16 | 7 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 9 | 40 | 13 | 14 | 2 | 4 | 0 | 0 | 0
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1 | 15 | 5 | 3 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will with hold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT02509494/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/94/NCT02509494/SAP_001.pdf